CLINICAL TRIAL: NCT06423508
Title: PRObing The Efficacy of Commercial Stage Storage Buffers and Evaluating Gut Metaproteome Variability Between Individuals
Acronym: PROTEGI
Status: Recruiting | Type: Observational
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Giacomo Carta, Postdoc, University of Vienna
Other Study IDs: EK_01149_3/05/2024
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Gut Microbiome; Buffer; Methodology Study; Fecal Microbiota; Variability
Keywords: storage buffer; fecal samples; human gut microbiome; metaproteomics; intra-individual variability; inter-individual variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- storage buffer standardisation: Identifying the most effective storage buffer for preserving protein integrity during the transportation of fecal samples from collection to processing sites, is essential for establishing consistent sample collection protocols, particularly for large-scale human fecal proteomic studies. Achieving consistency in sample collection is crucial for enabling individuals to have their gut health assessed via metaproteomics, unlocking the potential for personalized medicine and therapeutic interventions based on microbial communities.
- inter- and intra-individual variability: the aim is to explore the inter- and intra-individual variability observed in gut microbiome composition and functions from a proteomic perspective. Understanding inter-individual variability differences is crucial for personalized medicine. Recognizing and characterizing intra-individual variability is essential for accurately interpreting research findings, particularly in longitudinal studies or clinical monitoring scenarios. This study aims to elucidate these variabilities using proteomic data from volunteers' fecal samples, shedding light on the variables detected in the gut microbiome and providing insights into its dynamic nature

SUMMARY:
The study aims to assess the effectiveness of various commercial and non-hazardous buffers for the storage of human gut fecal samples over time. This evaluation will be conducted by comparing the performance of these buffers against directly frozen samples using metaproteomic analysis. The study is motivated by the need for standardized protocols for sample preservation in metaproteomic research, particularly focusing on protein preservation in fecal samples. By investigating proteomic, taxonomic, and functional identifications, the research seeks to provide insights into the reliability of these buffers as storage solutions. Additionally, the study plans to explore inter- and intra-individual variabilities at the proteome level by periodically collecting fecal samples from volunteers, complementing existing knowledge in metaproteomics. Overall, the study addresses a critical gap in the field and has the potential to enhance reproducibility and comparability across metaproteomic studies

DETAILED DESCRIPTION:
A. Introduction:

Metaproteomics studies the entire protein complement of a microbial community and offers insight into intricate ecosystems like the gut microbiome. Metaproteomics allows researchers to delve deep into gut microbiomes, providing insights into these microbial inhabitants, abundance and functional activities. This knowledge has been instrumental in elucidating the mechanisms underlying various diseases, such as inflammatory bowel disease, and obesity. Researchers can develop targeted strategies for personalized medicine and precision healthcare based on the underlying biology by identifying key protein signatures.

In gut microbiome studies, standardized sample collection and preservation are particularly crucial to preserve the integrity of the microbial community and its proteome. Indeed, to obtain reliable results it must be considered the susceptibility to environmental influences like temperature and oxygen amount. For gut microbiome metaproteomic studies, non-invasive or minimally invasive methods are preferred to minimize disruption, or contamination, and preserve the native microbial composition and protein profiles. Also, the sample handling and storage strategies affect the degradation of proteins and the microbial population stability. For this reason, immediate freezing, or preservation at low temperatures (e.g., -80°C) is often recommended to maintain sample integrity until analysis. However, using a cold chain for storage and transportation is not compatible with an on-site sampling strategy that is necessary for large-scale and delocalized studies. Moreover, it is less ideal, more expensive, and logistically tedious than potential room temperature options.

Furthermore, present knowledge of the fecal sample collection/preservation methods is based on preserving nucleic acids or metabolites during the transportation to the laboratory for analysis. However, protein preservation requires different strategies and studies are scarce and rely on adopting the devices or reagents used in the case of nucleic acids or metabolites analysis. Thus, tailored, and standardized protocols together with metadata collection are essential for ensuring reproducibility and comparability across metaproteomic studies.

The present study aims to evaluate the fitness of several commercial and non-hazardous buffers for the storage of human gut fecal samples over time. Fecal samples will be stored in five different buffers and will be benchmarked with directly frozen samples. Using metaproteomics the investigators will compare the proteomic, taxonomic, and functional identifications to understand the potential of these buffers as a reliable storage solution for human feces. This research is unique and to the best of our knowledge, no similar study has addressed this demanding question.

Preliminary evidence in humans has shown inter- and intra-individual variability of the proteomes of the host and microbiomes. In particular, the intra-individual taxonomic and functional variation in the gut microbiome seems to be lower than inter-individual variation over time. However, metatranscriptomics profiles exhibited comparable variability within and between subjects. Therefore, using metaproteomics, investigators aim to assess the inter- and intra-individual variabilities at the proteome level by studying fecal samples periodically collected from participants.

B. The academic and social relevance:

The first part of the study aims to define the most effective storage buffer for preserving protein integrity during sample transportation from the site of collection to the site of processing - a key factor in the future of metaproteomics applied to health and disease. Despite its importance, a similar evaluation has not been performed for proteomic applications. This knowledge will be critical for academic purposes to be used for large-scale human fecal proteomic studies. For people to have their gut health examined through metaproteomics and unlock the potential of microbial communities-based personalized medicine and therapeutic interventions there will be a requirement for consistent sample collection and this study will provide it.

The second part of the study is designed to understand the variability that can be observed in the gut microbiome composition and functions from the proteomics perspective. The gut microbiome is dynamic and is known to be altered by multiple factors such as diet, age, genetics, environment, etc. These variations can be broadly classified into inter- and intra-individual. Inter-individual variability refers to the differences observed between individuals within a population or group, and they can encompass a wide range of characteristics, including genetic makeup, physiological parameters, lifestyle factors, and environmental exposures. Understanding inter-individual variability from people of the same "community" is essential in fields such as personalized medicine, where tailored interventions account for individual differences to optimize treatment outcomes. Intra-individual variability, on the other hand, refers to variations observed within the same individual over time or under different conditions and can arise from biological fluctuations, such as circadian rhythms, hormonal fluctuations, or physiological responses to stimuli. Recognizing and characterizing intra-individual variability is crucial for accurately interpreting research findings and assessing the reliability of biological measurements, particularly in longitudinal studies or clinical monitoring scenarios. This study aims to understand these variabilities through the proteomics data collected from participants' fecal samples and define the variables detected in the gut microbiome.

C. Objectives:

1. To identify the effect of five different buffers used for the storage and transportation of collected human fecal material, by metaproteomic profiles.
2. To determine the variability in microbiota and host proteomes at the inter- and intra-individual levels.

D. Study Design:

For the first phase, the investigators will deploy the following protocol for on-site fecal sampling and transport preservation: The participants (recruited among the members of our laboratory/Division) will be provided with 18 tubes (numbered 1-18; 15 ml conical centrifuge tubes; Ref# 339650, Thermo Scientific and 18 easy-to-use commercial swabs (C1052-50, Zymo Research) or spatulas (DNAGenotek). The 18 tubes correspond to three storage time points of 6 different experimental conditions: an empty tube (without preservation liquid) as a control sample and 5 different non-hazardous fecal preservation liquids: (a) In-house buffer (called LB) with SDS and Urea, commercially obtained (b) Zymo DNA/RNA Shield (R1100, Zymo Research), (c) Copan Amies buffer (480CE, Copan Italia SpA), (d) OMNIgene•GUT (OM200, DNAGenotek), (e) OMNImet•GUT (ME200, DNAGenotek). Briefly, LB, Zymo Shield, and OM200 are known to contain detergents that help to preserve the biomolecules, Copan Amies buffer is a nutrient-free media known to keep the cells viable and shown to have applications in culturomics, and ME200 is solvent based useful in metabolomic applications. In addition, the participants will receive a commercial stool catcher that is displayed over the toilet for facilitating fecal sampling (Servoprax Stuhlfaenger, Reference number H7 61000-50 from www.medundorg.de) and a little box with ice packs in which the three Control samples will be stored and transported to the lab. These ice-stored Control samples are key to evaluating the performance of the different storage buffers. The participants will bring the samples to our laboratory in the following 24 hours. Upon reception in the lab, the Control samples will be stored at -80°C until further biochemical processing using established protocols. The rest of the samples will be stored at +20°C inside an orbital shaker incubator for a total of 2, 5, and 10 days (simulating different storage/transport times, thereof). At the end of these time points, the samples will be stored at -80°C until further biochemical processing using established protocols. The metaproteomic profiles (indicating the taxonomical and functional changes in the gut microbiome and the host physiology; as in the previous experiment from these samples will inform us about the best preservation liquid (defined as the one where the microbiome composition and function are more like the Control sample). This experiment is necessary for initiating Phase II of the study, and it is novel in the field as no guidelines are established for best in-house fecal sampling practices in metaproteomics. Six healthy participants (among the members of the Systems Biology of Pain laboratory, Division of Pharmacology & Toxicology, Department of Pharmaceutical Sciences) will be recruited. This is a randomized study with no participant groups. Samples will be collected once and distributed to 18 tubes representing different conditions. A sample size of 6 subjects will be enough to find the best preservation solution and the sampling will be performed one time under normal bowel movement by the participants. In addition, the participants will fill out a questionnaire (attached) that includes information like age, sex, Body Mass Index, the gastrointestinal symptoms rating scale (GSRS), administration of antibiotics in the last 30 days before sample collection, the Bristol stool form scale (BSFS), and the approximate time needed for sample collection in the 18 tubes (to account for potential effects due to oxidation processes).

For the second phase, the participants will be expected to collect fecal samples for 4 weeks during their regular defecation (ten different times maximum). They will be provided with an adequate number of 15ml conical centrifuge tubes (339650, Thermo Scientific) containing the best-performing preservation buffer (as defined in the first phase of the study, see above), and a commercial collection device with a stool catcher. Upon reception in the lab, the samples will be stored at -80°C until further biochemical processing using established protocols. In addition, the participants will fill out a questionnaire (see above). Participants will take part voluntarily in the experiment after receiving an explanation of all the risks and benefits of participating in the present study, and after signing the written informed consent form according to the Declaration of Helsinki (see the consent form, attached). The participants will be instructed and provided with necessary sampling devices to collect stool samples (see above) and submit the samples to the Department of Pharmacology and Toxicology at the earliest opportunity. Participants will be expected to complete self-administered questionnaires that include information like the one described above. For the second phase, 46 healthy participants (among the members of our laboratory/Division) will be recruited from both sexes (23 males and females) considering a possible dropout rate of 20%. This is a randomized study with no participant groups. The sample size was calculated based on the threshold of Eggerthella estimates with time. The statistics procedure used is F tests - two-way ANOVA with repeated measures with the following values Cohens'd = 0.75, 1-β= 0.80, and α= 0.05. A total of 400 - 460 samples are expected to be collected.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate after signing the informed consent form and
* being 18-70 years old.

Exclusion Criteria:

* take antibiotics during the previous 1 month
* had undergone gastrointestinal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers (among the members of our laboratory/Division) will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Eggerthella abundance | From enrollment to the end of treatment at 4 weeks
  Eggerthella abundance will be checked in to the Metaproteomic profile of each fecal samples and inter/intra-individual variability will be assessed

SECONDARY OUTCOMES:
Age | From enrollment to the end of treatment at 4 weeks
  Age will be collected from each participant during the first interview
Sex | From enrollment to the end of treatment at 4 weeks
  Sex will be collected from each participant during the first interview
Body Mass Index (BMI) | From enrollment to the end of treatment at 4 weeks
  BMI will be collected from each participant during the first interview
Antibiotic use | From enrollment to the end of treatment at 4 weeks
  Antibiotic use in the previous 1 month before the study enrollment, will be collected from each participant during the first interview
Bristrol Stool Form Scale (BSFS) | From enrollment to the end of treatment at 4 weeks
  The Bristol Stool Form Scale (BSFS), or Bristol stool scale, is a chart that can help classify stools into seven groups. Characterizing the stool based on its consistency can help identify if it is a healthy bowel movement. It will be administerd refearring to the the day(s) of the fecal sample collection(s)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, PhD, Principal Investigator — University of Vienna
Locations (1):
- UVienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
anonymized data will be provided under scientific plausible request sent by email to the principal investigator

REFERENCES:
- [Background] Gomez-Varela D, Xian F, Grundtner S, Sondermann JR, Carta G, Schmidt M. Increasing taxonomic and functional characterization of host-microbiome interactions by DIA-PASEF metaproteomics. Front Microbiol. 2023 Oct 16;14:1258703. doi: 10.3389/fmicb.2023.1258703. eCollection 2023. PMID 37908546